CLINICAL TRIAL: NCT07338188
Title: Optimization of the Perioperative Pathway Coordinated Through the Collection of Patient-reported Outcome Measures in Patients With Complex Care Needs: An Open-label Randomized Controlled Trial
Brief Title: PROMs-guided Perioperative Care in Patients With Complex Care Needs: An Open-label Randomized Controlled Trial
Acronym: OPTICAIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9965; 2025-A02288-41 (Other: N° IDRCB)
Record Dates: First submitted 2025-12-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Follow-up
Keywords: perioperative; surgery; Patient Reported Outcomes Mesuares (PROMs); Complex clinical situation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group In addition to routine follow up by the perioperative team including the surgical team, dedicated nurses will conduct PROMs based patients interviews. These interviews are carried out systematically and in a standardized manner during pre-hospitalization on postoperative days 1, 3, 14, 28 During the interview they will assist the patient with completing the QoR-15 questionnaire, allowing a snapshot of the patient's health status.
  If the nurse perceive an alteration of the patient healthstatus based on the interview, the patient may be refered to another healthcare professional (eg : surgeons, anesthesiologist, primary care physician for exemple) Preoperative contact by a nurse practitioner (NP) or registered nurse (RN) specialized in PROMs-based follow-up, and organization of perioperative follow-up on postoperative days 1, 3, 14, and 28.
  Interventions: Other: Patient-Reported Outcomes-based perioperative follow-up (QoR-15 focus)
- Control group (Active Comparator): follow-up by the perioperative team including the surgical team without the intervention of the dedicated PROMs based interviews team.
  Control groupe :
  The control group, on the other hand, will receive standard follow-up coordinated by the surgeon and in collaboration with the primary care physician and other community healthcare professionals, without intervention by a nurse practitioner (NP) or registered nurse (RN) and without PROMs-based follow-up.
  Interventions: Other: Patient-Reported Outcomes-based perioperative follow-up (QoR-15 focus)

INTERVENTIONS:
Other: Patient-Reported Outcomes-based perioperative follow-up (QoR-15 focus) — Description - Patient-Reported Outcomes-based perioperative follow-up (QoR-15 focus) The Patient-Reported Outcomes-based perioperative follow-up is a patient-centered approach that evaluates postoperative recovery using standardized questionnaires completed directly by the patient. This method highlights the patient's own perception of recovery-covering physical comfort, emotional state, independence, and pain control-rather than relying solely on clinical or physiological parameters.
  The Quality of Recovery-15 (QoR-15) questionnaire is a validated, short-form tool designed to measure the quality of postoperative recovery from the patient's perspective. It consists of 15 items covering five key dimensions:
  Physical comfort (pain, nausea, general well-being), Emotional state (anxiety, depression, feeling of support), Psychological support, Physical independence (ability to move or perform daily activities), Pain and symptom management.

SUMMARY:
This research aims to identify, as early as the preoperative phase, groups of patients likely to experience maximum clinical improvement through structured paramedical follow-up based on PROMs. However, the high heterogeneity of the included patients could have masked more pronounced effects in certain subgroups, particularly those at higher risk. Relying on a multicenter approach and a subgroup analysis, our study hypothesizes that certain patient profiles are more likely to significantly benefit from personalized follow-up based on PROMs. The objective is to validate the hypothesis that support through PROMs for patients in complex situations could allow for a more pronounced clinical effect. This follow-up will enable better targeting of interventions from the preoperative phase, optimize the use of healthcare resources, and improve quality, safety, and efficiency of perioperative pathways.

DETAILED DESCRIPTION:
The study is an open-label, multicenter, randomized controlled trial comparing two groups:

* A control group receiving the usual conventional follow-up, notably by the surgeon and the attending physician.
* An experimental group receiving, in addition to the usual conventional follow-up, follow-up by dedicated nurses focusing on the patient's perspective regarding their health status (OPTIMISTE follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Adult patient, with no upper age limit
* Undergoing scheduled or unscheduled surgery in a center participating in the research
* Presenting a care situation identified as complex, defined by a COMID score > 9
* Subject affiliated to a social health insurance scheme
* Subject able to understand the objectives and risks related to the research and to give informed consent, dated and signed

Exclusion Criteria:

* Inability to administer the mQoR-15f questionnaire (cognitive disorders, language barrier)
* Inability to provide the subject with informed information (subject in an emergency situation, difficulties in understanding, etc.)
* Patient who has already received previous follow-up by the OPTIMISTE team
* Patient enrolled in a therapeutic trial that may affect post-operative recovery quality
* Subject under legal protection, guardianship or curatorship
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-03-03 (Estimated); Study Completion 2028-04-03 (Estimated)

PRIMARY OUTCOMES:
The main objective is to evaluate the effectiveness of a perioperative follow-up integrating the patient's perspective based on their perceived health status. | Between the baseline consultation and "day 35"
  Evolution of a modified version of the French Quality-Of-Recovery 15 score (QoR-15f) between the baseline consultation and postoperative "day 35" (depending on the groups: with or without the OPTISMISTE program).
  The evoluation is scored from 0 to 150 (A higher score indicates better quality of recovery.)